CLINICAL TRIAL: NCT01296906
Title: Population Versus Practice-based Interventions to Increase Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 10-0823; 1RC1LM010513-01 (NIH)
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Health Services Research; Comparative Effectiveness; Immunization
Keywords: Reminder/recall messages; reminders; recall; immunizations; immunization information systems; effectiveness of reminder/recall; population-based reminder/recall

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Population-based Reminder/Recall (Experimental): Recall is performed centrally by public health departments for all children in need of immunizations in a geographic area.
  Interventions: Behavioral: Recall conducted centrally by local health department
- Practice-based Reminder/Recall (Experimental): Reminder/Recall is performed by individual private practices for their patients who appear in need of immunizations.
  Interventions: Behavioral: Recall conducted by private practices

INTERVENTIONS:
Behavioral: Recall conducted by private practices — All practices in these counties will receive training on practice-based R/R using the Colorado Immunization Information System (CIIS or immunization registry). Practices will receive a recommended schedule for conducting recall in 19-35 month children and educational materials to use within their practices to promote compliance with the infant vaccination schedule. Individual practices will make their own decisions about the extent to which they follow the recommendations and implement recall within their practice. Although the study team will not provide them with any additional interventions, we will track any other interventions they independently do (websites, newsletters, telephone informational systems) in order to assess the effect of these additional interventions.
  Arms: Practice-based Reminder/Recall
Behavioral: Recall conducted centrally by local health department — A centralized recall of children 19-35 months will be conducted through local health departments. CIIS will identify a cohort of 19-35 month olds with an who are in need of an immunization and will coordinate up to 3 mailers to children who are not current for recommended immunizations.
  Arms: Population-based Reminder/Recall

SUMMARY:
One of the nation's major health priorities, as outlined in Healthy People 2010, is to increase the proportion of children aged 19 to 35 months who have received all universally recommended vaccines. This study will compare two interventions for increasing immunization rates in this age group, one using well-studied primary care practice-based methods and the other using innovative technologies to increase immunization rates at the population-level. Results of this study will provide data that will be relevant nationally in guiding future investment of resources to increase up-to-date rates in young children prior to school entry.

Hypothesis: Population-based approaches will be more effective than practice-based interventions at increasing immunizations among 19-35 month olds.

ELIGIBILITY:
Inclusion Criteria:

* child between the age of 19-35 months
* has an address in a specified study county in the state immunization registry
* child is in need of at least one recommended immunization

Exclusion Criteria:

* child has opted out of the state immunization registry
* child is up-to-date on all recommended immunizations

Min Age: 19 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31567 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluate effectiveness of population-based reminder/recall methods versus practice-based reminder/recall methods in 14 Colorado counties (rural and urban) | 6 months post-intervention (December 2010)
  The primary outcome measures will be: 1) change in up-to-date rates from baseline levels 6 months after the intervention (T-1) for 19-35 month olds in population-based compared to practice-based intervention counties and 2) percent of children who were not up-to-date prior to recall (T-0) who received any additional new vaccine in each type of intervention county.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver, Colorado, United States

REFERENCES:
- [Background] Briss PA, Rodewald LE, Hinman AR, Shefer AM, Strikas RA, Bernier RR, Carande-Kulis VG, Yusuf HR, Ndiaye SM, Williams SM. Reviews of evidence regarding interventions to improve vaccination coverage in children, adolescents, and adults. The Task Force on Community Preventive Services. Am J Prev Med. 2000 Jan;18(1 Suppl):97-140. doi: 10.1016/s0749-3797(99)00118-x. PMID 10806982
- [Background] Recommendations regarding interventions to improve vaccination coverage in children, adolescents, and adults. Task Force on Community Preventive Services. Am J Prev Med. 2000 Jan;18(1 Suppl):92-6. No abstract available. PMID 10806981
- [Background] Tierney CD, Yusuf H, McMahon SR, Rusinak D, O' Brien MA, Massoudi MS, Lieu TA. Adoption of reminder and recall messages for immunizations by pediatricians and public health clinics. Pediatrics. 2003 Nov;112(5):1076-82. doi: 10.1542/peds.112.5.1076. PMID 14595049
- [Background] Murray DM, Varnell SP, Blitstein JL. Design and analysis of group-randomized trials: a review of recent methodological developments. Am J Public Health. 2004 Mar;94(3):423-32. doi: 10.2105/ajph.94.3.423. PMID 14998806
- [Derived] Kempe A, Saville A, Dickinson LM, Eisert S, Reynolds J, Herrero D, Beaty B, Albright K, Dibert E, Koehler V, Lockhart S, Calonge N. Population-based versus practice-based recall for childhood immunizations: a randomized controlled comparative effectiveness trial. Am J Public Health. 2013 Jun;103(6):1116-23. doi: 10.2105/AJPH.2012.301035. Epub 2012 Dec 13. PMID 23237154